CLINICAL TRIAL: NCT05553639
Title: A Phase 1/2 Study of Replicating Arenavirus-based Vector(s) Encoding Prostate Cancer-Associated Antigens in Participants With Metastatic Castration-Resistant Prostate Cancer
Brief Title: HB-302/HB-301 Therapy in Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Decision by the company to terminate the H-300-001 study early for non-safety related reasons.
Sponsor: Hookipa Biotech GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-300-001
Record Dates: First submitted 2022-08-17; First posted 2022-09-23 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer Metastatic
Keywords: Prostate; Prostate Cancer; Metastatic; Metastatic Cancer; Metastatic Prostate Cancer; Castration Resistant; Castration Resistant Prostate Cancer; mCRPC; CRPC; Vaccine; Viral Vector; Viral Therapy; Immunotherapy; Vaccine Therapy
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HB-302/HB-301 Alternating 2-Vector Therapy Intravenously (IV) (Experimental): HB-302/HB-301 Alternating 2-Vector Therapy Intravenously (IV)
  Interventions: Biological: HB-302/HB-301 Alternating 2-Vector Therapy

INTERVENTIONS:
Biological: HB-302/HB-301 Alternating 2-Vector Therapy — Alternating Therapy of HB-302 and HB-301. The first 5 doses will be administered every 3 weeks. The 6th dose will be administered 6 weeks after the 5th dose. Subsequent doses will be administered every 6 weeks.

SUMMARY:
This is a first-in-human Phase 1/2, multinational, multicenter, open-label study of HB-302/HB-301 alternating 2-vector therapy in participants with metastatic castration-resistant prostate cancer (mCRPC) comprising 2 phases: a Phase 1 Dose Escalation and recommended Phase 2 dose (RP2D) Confirmation, and a Phase 2 Dose Expansion.

DETAILED DESCRIPTION:
This is a first-in-human Phase 1/2, multinational, multicenter, open-label study of HB-302/HB-301 alternating 2-vector therapy in participants with metastatic castration-resistant prostate cancer (mCRPC) comprising 2 phases: a Phase 1 Dose Escalation and recommended Phase 2 dose (RP2D) Confirmation, and a Phase 2 Dose Expansion.

The Phase 1 Dose Escalation will evaluate HB-302/HB-301 alternating 2-vector therapy for safety and tolerability, preliminary efficacy and immunogenicity, and determination of a safe recommended Phase 2 dose (RP2D). A confirmatory cohort (or cohorts) will inform the determination of the RP2D. The Phase 2 Dose Expansion will assess HB-302/HB-301 alternating 2-vector therapy at the RP2D defined in the Phase 1 part of the study.

Study drugs HB-301 and HB-302 are genetically-engineered replicating vectors based on the arenavirus lymphocytic choriomeningitis virus (LCMV) and arenavirus Pichinde virus (PICV), respectively. HB-301 and HB-302 express the same transgenes encoding 2 prostate cancer-associated antigens: prostatic acid phosphatase (PAP) and prostate specific antigen (PSA). HB-302/HB-301 Alternating 2-vector therapy will be administered intravenously every 3 weeks (Q3W) for the first 5 doses and every 6 weeks (Q6W) from the fifth dose and onward. HB-302 is to be administered first followed 3 or 6 weeks later by HB-301.

In total, approximately 70 participants aged 18 years and older will be enrolled in this study to receive HB-302/HB-301 alternating 2-vector therapy.

About 40 Investigators and study sites in the United States (US) and Europe are expected to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants ≥18 years of age on day of signing the informed consent form (ICF)
2. Confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features, and evidence of metastatic disease.
3. Documented castration-resistant disease with serum level of testosterone <50 ng/dL (1.7 nmol/L).
4. Have been treated with at least one second-generation androgen receptor signaling inhibitor (ARSI) (e.g., enzalutamide)

   * No prior chemotherapy regimens are permitted (docetaxel in the castration-sensitive setting is acceptable)
   * Participants must have had disease progression on SOC therapy assessed by the Investigator.
   * Antiandrogen/ARSI withdrawal must take place at least 2 weeks before enrollment unless agreed otherwise between the Sponsor and the Investigator. LHRH agonists or antagonists should be continued.
5. Must have ≥1 metastatic lesion that is present on baseline imaging

   * Participants with liver metastasis are not eligible to enroll in this study
   * Participants with only bone metastasis present at baseline are eligible to enroll in this study
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 1.
7. Prior curative radiation therapy must have been completed at least 4 weeks prior to study drug administration. Prior focal palliative radiotherapy must have been completed at least 2 weeks prior to study drug administration.
8. Screening laboratory values must meet the criteria for adequate organ function that will be decided by the investigator.

Exclusion Criteria:

1. Any serious or uncontrolled medical disorder that, in the opinion of the Investigator, may increase the risk associated with study participation or study treatment administration, impair the ability of the participant to receive study treatment, or interfere with the interpretation of the study results. This includes clinically significant (i.e., active) cardiovascular disease, including cerebral vascular accident/stroke and myocardial infarction less than 6 months prior to enrollment, unstable angina, congestive heart failure (New York Heart Association Classification Class II), or serious uncontrolled cardiac arrhythmias (including prolonged corrected QT interval, uncontrolled atrial fibrillation, etc.)
2. Uncontrolled pain or uncontrolled symptoms related to worsening of underlying disease or symptomatic bone metastasis.
3. An active autoimmune disease that has required systemic treatment in past 2 years.

   • Note: Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed.
4. Has received the following immunosuppressive or systemic replacement medication:

   * Immunosuppressive doses of systemic medication, such as steroids or absorbed topical steroids (doses >10 mg/day prednisone or equivalent), within 14 days of the first administration of study treatment.

     • Note: inhaled or topical steroids and adrenal replacement in doses equivalent to >10 mg/day prednisone are permitted in the absence of active autoimmune disease.
   * Any chronic immunosuppressive medication within 6 months prior to the first administration of study treatment (unless agreed otherwise between the Sponsor and the Investigator on a case-by-case basis).
5. Has received a live or live-attenuated vaccine within 30 days of planned start of study therapy, unless agreed otherwise between the Sponsor and Investigator.

   • Administration of non-live vaccines is allowed.
6. Currently participating in or has participated in a study of an investigational agent or has used an investigational device treatment, within 4 weeks prior to the first dose of treatment.
7. Allogeneic tissue/solid organ transplant (e.g., allogeneic stem cell transplantation, xenogeneic transplant).
8. Active central nervous system (CNS) metastases and/or carcinomatous meningitis and/or epidural or neurological metastasis.
9. Active infection requiring systemic therapy.
10. Positive COVID-19 test in 6 weeks prior to the enrollment.
11. Known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
12. Known history of Hepatitis B (HBV) (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C (HCV) infection (defined as HCV ribonucleic acid [RNA] is detected [qualitative]).
13. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All participants will be male.
Enrollment: 12 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2024-04-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Phase I | 1. First 42 days of treatment, 2. Approximately 6 months
  1. Frequency and type of DLT. A DLT is defined as an adverse event that is unrelated to disease progression, intercurrent illness, or concomitant medications and is occurring during the first 42 days of treatment.
  2. Frequency and severity of adverse events (AEs). Using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grading scale, version 4.0.
Phase II | Up to 2 years
  The number of the participants with preliminary anti-tumor activity defined as:
  - Objective Response Rate (ORR) per RECIST v1.1/iRECIST criteria

SECONDARY OUTCOMES:
Phase I | Approximately 2 years
  Number of participants with an antitumor response. According to the chosen RECIST and PCWG3 criteria including PSA decline.
Phase II | Up to 24 months
  1. The number of participants with preliminary anti-tumor activity. According to the chosen RECIST and PCWG3 criteria including PSA decline.
  2. Frequency and severity of adverse events (AEs). Using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) grading scale, version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Development, Study Director — Hookipa Biotech GmbH
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - California Cancer Associates for Research & Excellence (cCARE), San Marcos, California
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Emory University Hospital, Atlanta, Georgia
  - The Cancer Institute of New Jersey CINJ Rutgers, New Brunswick, New Jersey
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Providence Cancer Institute, Portland, Oregon
  - Thompson Cancer Survival Center, Knoxville, Tennessee